CLINICAL TRIAL: NCT00613626
Title: A Randomized Double Blind Phase II Trial of Cisplatin Plus Etoposide With/Without Concurrent ZD6474 in Patients With Previously Untreated Extensive Stage Small Cell Lung Cancer: Hoosier Oncology Group LUN06-113
Brief Title: Cisplatin + Etoposide +/- Concurrent ZD6474 in Previously Untreated Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUN06-113
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Extensive Stage; Untreated
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin; Etoposide; vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: ZD6474 Matched Placebo (Placebo Comparator): Subjects will receive cisplatin 60 mg/m2 IV day 1 plus etoposide 120 mg/m2 IV days 1, 2, and 3 every 21 days for a total of 4 cycles plus ZD6474 matched placebo oral daily to be continued for the duration of the study. Prophylactic antiemetics will be given at the discretion of the treating investigator.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: Placebo
- Arm B: ZD6474 (Active Comparator): Subjects will receive cisplatin 60 mg/m2 IV day 1 plus etoposide 120 mg/m2 IV days 1, 2, and 3 every 21 days for a total of 4 cycles plus ZD6474 100mg oral daily to be continued for the duration of the study. Prophylactic antiemetics will be given at the discretion of the treating investigator.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: ZD6474
- Safety Lead-In (Experimental): Subjects will receive cisplatin 60 mg/m2 IV day 1 plus etoposide 120 mg/m2 IV days 1, 2, and 3 every 21 days for a total of 4 cycles plus ZD6474 100mg oral daily to be continued for the duration of the study. Prophylactic antiemetics will be given at the discretion of the treating investigator. The safety lead-in will be conducted to determine the safety of the combination of ZD6474 and cisplation + etopiside. If this combination is found to be unsafe, no patients will be randomized in the Phase II portion of the trial. If the combination is deemed safe according to the protocol, participants from the safety lead-in cohort will not be included in the efficacy analysis.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: ZD6474

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 60 mg/m2 IV day 1 every 21 days for a total of 4 cycles
Drug: Etoposide — Etoposide 120 mg/m2 IV days 1, 2, and 3 every 21 days for a total of 4 cycles
Drug: Placebo — Matched placebo oral daily
  Arms: Arm A: ZD6474 Matched Placebo
Drug: ZD6474 — ZD6474 100mg oral daily to be continued for the duration of the study.
  Arms: Arm B: ZD6474; Safety Lead-In

SUMMARY:
At this point in the treatment of extensive stage SCLC, we have reached a plateau in survival with conventional chemotherapy and newer regimens are greatly needed. It has been noted that patients with increased VEGF levels have a poorer prognosis. Anti-angiogenic agents hold significant promise in the treatment of patients with extensive stage SCLC. ZD6474, a new inhibitor of the VEGFR-2, has shown favorable action in NSCLC.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Arm A:

Cisplatin 60mg/m2 Day 1 + Etoposide 120mg/m2 Day 1,2,3 + Placebo oral daily given continuously for the duration of the study

Arm B:

Cisplatin 60mg/m2 Day 1 + Etoposide 120mg/m2 Day 1,2,3 + ZD6474 100mg oral daily given continuously for the duration of the study

For both arms, PE and toxicity evaluation prior to each cycle and disease assessment by imaging every 2 cycles. Patients with non-PD and acceptable toxicity will continue protocol therapy; patients with progressive disease or excessive toxicity will be taken off treatment. Cycles will be repeated every 21 days up to a total of 4 cycles.

ECOG Performance Status of 0 or 1

Life Expectancy: Not specified

Hematopoietic:

* Platelets > 100K/mm3
* Absolute neutrophil count (ANC) > 1.5K/mm3

Hepatic:

* Bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST) < 2.5 x ULN or < 5 x ULN if judged by the investigator to be related to liver metastases
* Alkaline phosphatase < 2.5 x ULN or < 5 x ULN if judged by the investigator to be related to liver metastases

Renal:

* Serum creatinine < 1.5 x ULN or Calculated creatinine clearance of > 45 cc/min using the Cockcroft-Gault formula

Cardiovascular:

* No clinically significant cardiac event such as myocardial infarction; New York Heart Association (NYHA) classification of heart disease >2 (see SPM) within 3 months prior to registration for protocol therapy
* No presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
* No history of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is permitted.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of chemotherapy-naïve, extensive, small cell lung cancer.
* Measurable disease according to RECIST and obtained by imaging within 28 days prior to being registered for protocol therapy.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age 18 years or older at the time of consent.
* Potassium ≥4.0 mmol/L and <5.5mmol/L (supplementation is allowed).
* Calcium within normal range (supplementation is allowed).
* Magnesium within normal range (supplementation is allowed).

Exclusion Criteria:

* No prior EGFR inhibitor or antiangiogenic agent allowed.
* No prior hormonal therapy.
* No symptomatic brain metastasis.
* No clinically significant infections as judged by the treating investigator.
* No evidence of severe or uncontrolled other systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.
* No previous history of QTc prolongation as a result of medication that required discontinuation of that medication.
* No congenital long QT syndrome or known 1st degree relative with unexplained sudden death under 40 years of age.
* No presence of left bundle branch block (LBBB.)
* No QTc with Bazett's correction that is unmeasurable, or ≥480 msec on screening ECG obtained within 7 days prior to registration for protocol therapy. If a subject has QTc ≥480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be <480 msec in order for the subject to be eligible for the study.
* No concomitant (within 14 days prior to registration for and during protocol therapy) medication associated with Torsades de Pointes or cause QTc prolongation, is allowed. Medications that prolong QT, but are not strictly associated with Torsades, are allowed if medically necessary and will require increased ECG and electrolyte monitoring.
* No uncontrolled hypertension (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg).
* No currently active diarrhea that may affect the ability to absorb ZD6474.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, Gleason < grade 7 prostate cancers, or other cancer for which the subject has been disease-free for at least 5 years.
* Major surgery must be completed greater than 28 days prior to registration for protocol therapy and healed surgical incision is required.
* No concomitant (within 14 days prior to registration for and during protocol therapy) medications that are potent inducers (rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital and St. John's Wort) of CYP3A4 function.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 8 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.
* Females must not be breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Oncology Group, Inc.
Locations (19):
- United States (19):
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - IN Onc/Hem Associates, Indianapolis, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital & Health Centers, Indianapolis, Indiana
  - IU Health Arnett Cancer Center, Lafayette, Indiana
  - Horizon Oncology Researcg, Lafayette, Indiana
  - IU Health at Ball Memorial Hospital, Muncie, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Methodist Cancer Center, Omaha, Nebraska
  - Hematology Oncology Associates S.J., P.A., Mount Holly, New Jersey
  - Providence Portland Medical Center, Portland, Oregon
  - Pennsylvania Oncology-Hematology Associates, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Rachel E. Sanborn, Jyoti D. Patel, Gregory A. Masters, Nagesh Jayaram, Anthony W. Stephens, Michael J. Guarino, Jamal Ghazi Misleh, Corinne E. Williams, Jingwei Wu, Nasser H. Hanna. A randomized double-blind phase II trial of platinum (P) plus etoposide (E) with or without concurrent ZD6474 (Z) in patients (pts) with previously untreated extensive-stage (ES) small cell lung cancer (SCLC): Hoosier Oncology Group LUN06-113. J Clin Oncol 32:5s, 2014 (suppl; abstr 7506)
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: ZD6474 Matched Placebo | Arm B: ZD6474 | Safety Lead-In
Started | 33 | 34 | 7 (These participants provided the toxicity data to determine if ZD6474+Etopiside+Cisplatin was safe.)
1st Dose ZD6474 | 33 | 34 | 7
Completed | 33 | 33 | 7
Not Completed | 0 | 1 | 0
Not completed — Ineligible | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects 18 years of age or older at time of consent, ECOG Performance Status of 0-1 14 days prior to registration, and histological or cytological proof of chemotherapy naive extensive small cell cancers or neuroendocrine cancers that are high grade or poorly differentiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: ZD6474 Matched Placebo | Arm B: ZD6474 | Safety Lead-In | Total
Number analyzed (Participants) | 33 | 33 | 7 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.58 (10.92) | 63.80 (5.90) | 66.14 (3.34) | 62.94 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 2 | 32
  Male | 17 | 19 | 5 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 29 | 7 | 67
  Unknown or Not Reported | 2 | 4 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 32 | 29 | 5 | 66
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 7 | 73
ECOG Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group Score
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  participants
    0 | 12 | 11 | 2 | 25
    1 | 21 | 22 | 5 | 48
Liver Metastases [Number; unit: participants]
  Present | 16 | 13 | 1 | 30
  Absent | 17 | 20 | 6 | 43
Brain Metastases [Number; unit: participants]
  Present | 10 | 10 | 5 | 25
  Absent | 23 | 23 | 2 | 48
Platinum Therapy [Number; unit: participants]
  Cisplatin | 17 | 17 | 7 | 41
  Carboplatin | 16 | 16 | 0 | 32

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression - Median Time to Progression and Log-Rank Test
Description: Kaplan-Meier analysis comparing arm A to arm B. Median time to progression and log-rank test. Safety lead-in participants are not included in this analysis per protocol.
Time Frame: 24 months
Population: Two participants from Arm A and Two Participants from Arm B were inevaluable for the time to disease progression analysis. (Reasons inevaluable include: toxicity and withdrawal of consent)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: ZD6474 Matched Placebo | Arm B: ZD6474
Number analyzed (Participants) | 31 | 31
Months | 5.68 [3.98 to 6.41] | 5.62 [5.09 to 6.24]
Statistical Analysis 1: Comparison: Arm A: ZD6474 Matched Placebo vs Arm B: ZD6474; A one-sided log rank test with an overall sample size of 68 subjects (of which 34 are in arm A and 34 are in arm B) achieves 80% power at a 0.10 significance level to detect a difference of 3 months in PFS between 4 month median PFS and 7 month median PFS; Test type: Superiority or Other; p = 0.10, Log Rank; Median Difference (Final Values) = 3, Standard Error of Mean 22.718
Statistical Analysis 2: Comparison: Arm A: ZD6474 Matched Placebo vs Arm B: ZD6474; Test type: Superiority or Other; p = 0.9518, Log Rank — P-Value (2-tailed) is calculated based on the unstratified log-rank test; Degrees of freedom=1

2. Secondary Outcome: Percentage of Participants With Grade 3/4 Hematologic and Non-Hematologic Toxicities
Description: Percentage of participants who experienced grade 3/4 hematologic and non-hematologic toxicities. Participants from Arm A were compared to subjects from Arm B + Safety Lead-In.
Time Frame: 6 weeks (2 Cycles)
Population: The participants from the safety run-in cohort were combined with the participants from ARM B for analysis of safety.
Measure: Number; unit: percentage of participants
Groups:
- Arm B: ZD6474 + Safety Lead-In: Subjects will receive cisplatin 60 mg/m2 IV day 1 plus etoposide 120 mg/m2 IV days 1, 2, and 3 every 21 days for a total of 4 cycles plus ZD6474 100mg oral daily to be continued for the duration of the study. Prophylactic antiemetics will be given at the discretion of the treating investigator.
  Cisplatin: Cisplatin 60 mg/m2 IV day 1 every 21 days for a total of 4 cycles
  Etoposide: Etoposide 120 mg/m2 IV days 1, 2, and 3 every 21 days for a total of 4 cycles
  ZD6474: ZD6474 100mg oral daily to be continued for the duration of the study.
Arm/Group | Arm A: ZD6474 Matched Placebo | Arm B: ZD6474 + Safety Lead-In
Number analyzed (Participants) | 33 | 40
percentage of participants
  Grade 3/4 Hematologic Toxicity | 11.00 | 13.75
  Grade 3/4 Non-Hematologic Toxicity | 2.71 | 4.30

3. Secondary Outcome: Measure the Response Rate (CR + PR) in Each Arm
Description: Response assessments completed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST Therasse et al., 2000). Complete Response (CR) is defined as: Disappearance of all target lesions. Partial Response (PR) is defined as: >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 24 months
Population: 12 participants are excluded due to missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: ZD6474 Matched Placebo | Arm B: ZD6474
Number analyzed (Participants) | 26 | 28
percentage of participants | 65.38 [47.10 to 83.67] | 50.00 [31.48 to 68.52]
Statistical Analysis 1: Comparison: Arm A: ZD6474 Matched Placebo vs Arm B: ZD6474; Test type: Superiority or Other; p = 0.2533, Difference in Rates; P-value (two-tailed) is calculated based on an unadjusted, normal-distribution approximation for the difference in rates

4. Secondary Outcome: Measure Disease Control Rate (CR + PR+ SD) in Each Arm
Description: Response assessments completed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST Therasse et al., 2000). Complete Response (CR) is defined as: Disappearance of all target lesions. Partial Response (PR) is defined as: >=30% decrease in the sum of the longest diameter of target lesions. Stable Disease (SD) is defined as: neither a partial response or progressive disease ( >=20% increase in the sum of the longest diameter of the target lesions).
Time Frame: 24 months
Population: 12 participants were not analyzed due to missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: ZD6474 Matched Placebo | Arm B: ZD6474
Number analyzed (Participants) | 26 | 28
percentage of participants | 73.08 [56.03 to 90.13] | 75.00 [58.96 to 91.04]
Statistical Analysis 1: Comparison: Arm A: ZD6474 Matched Placebo vs Arm B: ZD6474; Test type: Superiority or Other; p = 0.8720, Difference in Rates

5. Secondary Outcome: Measure Overall Survival for Each Arm
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: ZD6474 Matched Placebo | Arm B: ZD6474
Number analyzed (Participants) | 33 | 33
Months | 9.23 [6.64 to 11.27] | 13.24 [7.82 to 17.38]
Statistical Analysis 1: Comparison: Arm A: ZD6474 Matched Placebo vs Arm B: ZD6474; Test type: Superiority or Other; p = 0.4577, Log Rank

6. Secondary Outcome: Assess VEGF Polymorphisms and Correlate Subject Response
Time Frame: 24 months
Population: This data was not collected for the safety lead-in participants.
Measure: Number; unit: probability
Arm/Group | Arm A: ZD6474 Matched Placebo | Arm B: ZD6474
Number analyzed (Participants) | 33 | 33
probability
  Survival Analysis VEGF SNP rs699947 | 0.4642 | 0.6148
  Survival Analysis VEGF SNP rs3025039 | 0.1234 | 0.2050
  Survival Analysis VEGF SNP rs2019063 | 0.3968 | 0.8486
  Survival Analysis VEGF SNP rs1570360 | 0.0712 | 0.4426
  Survival Analysis VEGF SNP rs833061 | 0.4642 | 0.6148
  Response Analysis VEGF rs699947 | 0.6034 | 0.6034
  Response Analysis VEGF SNP rs3025039 | 0.1842 | 0.1842
  Response Analysis VEGF SNP rs2019063 | 0.0959 | 0.0959
  Response Analysis VEGF SNP rs1570360 | 0.4586 | 0.4586
  Response Analysis VEGF SNP rs833061 | 0.6034 | 0.6034
Statistical Analysis 1: Comparison: Arm A: ZD6474 Matched Placebo vs Arm B: ZD6474; Data was not collected for safety lead-in participants and these participants were not included in the analysis; Test type: Superiority or Other; Cox Proportional Hazard = 0.05 — Survival analysis of VEGF variants using cox proportional hazard analysis in arm A and arm B
Statistical Analysis 2: Comparison: Arm A: ZD6474 Matched Placebo vs Arm B: ZD6474; Test type: Superiority or Other; Logistic Regression Analysis = 0.05 — Objective Response Analysis of VEGF variants using Logistic Regression Analysis in arm A and arm B

ADVERSE EVENTS:
Arm/Group | Arm A: ZD6474 Matched Placebo | Arm B: ZD6474
Serious Adverse Events (participants affected / at risk) | 8/33 | 14/41
Other Adverse Events (participants affected / at risk) | 32/33 | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: ZD6474 Matched Placebo (N=33) | Arm B: ZD6474 (N=41)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ISCHEMIA/INFARCTION (Cardiac disorders) | 1 (1) | 2 (2)
CONFUSION (Nervous system disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 1 (1) | 1 (1)
HEMOGLOBIN (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
HEMORRHAGE, GI / LOWER GI NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / BRONCHOPULMONARY NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / ARTERY (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / BLADDER (URINARY) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1) | 1 (1)
INFECTION WITH UNKNOWN ANC / MEDIASTINUM NOS (Infections and infestations) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (2)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PAIN / BACK (General disorders) | 0 (0) | 1 (1)
PANCREATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
PLATELETS (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 0 (0) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: ZD6474 Matched Placebo (N=33) | Arm B: ZD6474 (N=41)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 5 (9) | 5 (5)
ALKALINE PHOSPHATASE (Investigations) | 5 (5) | 4 (5)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 0 (0) | 2 (2)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 3 (4) | 2 (2)
ANOREXIA (Gastrointestinal disorders) | 11 (12) | 13 (14)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 3 (4) | 1 (1)
BRONCHOSPASM, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Investigations) | 1 (1) | 1 (1)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 3 (6) | 6 (9)
CARDIAC ISCHEMIA/INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 4 (4) | 2 (2)
CONFUSION (Nervous system disorders) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 9 (12) | 9 (11)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 0 (0) | 1 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 12 (13)
CREATININE (Investigations) | 3 (3) | 7 (7)
CYSTITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 1 (1) | 4 (6)
DENTAL: TEETH (Gastrointestinal disorders) | 1 (1) | 1 (1)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 2 (2) | 9 (10)
DIZZINESS (Nervous system disorders) | 2 (8) | 5 (5)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 (1) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 0 (0) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 18 (22) | 19 (21)
EDEMA: HEAD AND NECK (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
EDEMA: LIMB (Blood and lymphatic system disorders) | 8 (12) | 2 (2)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 24 (33) | 26 (36)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 3 (3) | 2 (2)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
FLUSHING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
GASTRITIS (INCLUDING BILE REFLUX GASTRITIS) (Gastrointestinal disorders) | 1 (1) | 0 (0)
GLAUCOMA (Eye disorders) | 1 (1) | 0 (0)
GLOMERULAR FILTRATION RATE (Investigations) | 1 (1) | 0 (0)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 10 (12) | 9 (13)
GLUCOSE, SERUM-LOW (HYPOGLYCEMIA) (Investigations) | 0 (0) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 10 (13) | 12 (15)
HEARING: PATIENTS WITHOUT BASELINE AUDIOGRAM AND NOT ENROLLED IN A MONITORING PROGRAM (Ear and labyrinth disorders) | 2 (2) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 3 (3) | 6 (6)
HEMOGLOBIN (Blood and lymphatic system disorders) | 16 (31) | 14 (24)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
HEMORRHAGE, GI / UPPER GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / RESPIRATORY TRACT NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
HOT FLASHES/FLUSHES (Endocrine disorders) | 1 (2) | 0 (0)
HYPERTENSION (Cardiac disorders) | 6 (6) | 10 (16)
HYPOTENSION (Cardiac disorders) | 1 (1) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / MUCOSA (Infections and infestations) | 0 (0) | 1 (1)
INFECTIONWITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / PHARYNX (Infections and infestations) | 0 (0) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / UPPER AIRWAY NOS (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC / WOUND (Infections and infestations) | 0 (0) | 1 (1)
INSOMNIA (General disorders) | 6 (6) | 6 (6)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 7 (11) | 12 (20)
LIPASE (Investigations) | 0 (0) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 7 (11) | 12 (16)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
METABOLIC/LABORATORY - OTHER (SPECIFY, __) (Investigations) | 1 (1) | 0 (0)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 0 (0) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 7 (7) | 5 (5)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 4 (4) | 4 (4)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 3 (3) | 7 (8)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 0 (0) | 2 (2)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTRAOCULAR (Eye disorders) | 0 (0) | 2 (2)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (SPECIFY, __) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 14 (18) | 16 (17)
NEUROENDOCRINE: ADH SECRETION ABNORMALITY (E.G., SIADH OR LOW ADH) (Endocrine disorders) | 1 (1) | 0 (0)
NEUROPATHY: CRANIAL / CN V MOTOR-JAW MUSCLES; SENSORY-FACIAL (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY: MOTOR (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 4 (4) | 4 (4)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 11 (17) | 19 (26)
OPHTHALMOPLEGIA/DIPLOPIA (DOUBLE VISION) (Eye disorders) | 0 (0) | 1 (1)
OTITIS, MIDDLE EAR (NON-INFECTIOUS) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 4 (4) | 2 (2)
PAIN / BACK (General disorders) | 10 (10) | 8 (8)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN / BUTTOCK (General disorders) | 1 (1) | 1 (1)
PAIN / CARDIAC/HEART (Cardiac disorders) | 1 (1) | 0 (0)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7)
PAIN / DENTAL/TEETH/PERIDONTAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (5)
PAIN / FACE (General disorders) | 0 (0) | 1 (1)
PAIN / HEAD/HEADACHE (General disorders) | 6 (6) | 5 (7)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
PAIN / NECK (General disorders) | 4 (4) | 1 (1)
PAIN / ORAL CAVITY (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN / PAIN NOS (General disorders) | 1 (1) | 2 (2)
PAIN / PLEURA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PAIN / STOMACH (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN / THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PAIN - OTHER (SPECIFY, __) (General disorders) | 3 (3) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 3 (3)
PANCREATIC ENDOCRINE: GLUCOSE INTOLERANCE (Endocrine disorders) | 2 (2) | 0 (0)
PHOSPHATE, SERUM-LOW (HYPOPHOSPHATEMIA) (Investigations) | 2 (2) | 4 (4)
PLATELETS (Blood and lymphatic system disorders) | 5 (9) | 10 (11)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 3 (3) | 4 (4)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 5 (10) | 6 (7)
PROLONGED QTC INTERVAL (Cardiac disorders) | 1 (1) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 (3) | 8 (10)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
RASH: DERMATITIS ASSOCIATED WITH RADIATION / CHEMORADIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RIGORS/CHILLS (General disorders) | 0 (0) | 1 (1)
SODIUM, SERUM-HIGH (HYPERNATREMIA) (Investigations) | 1 (1) | 2 (2)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 8 (9) | 9 (11)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SWEATING (DIAPHORESIS) (General disorders) | 2 (2) | 2 (2)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 2 (2) | 2 (2)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1) | 1 (1)
THYROID FUNCTION, LOW (HYPOTHYROIDISM) (Endocrine disorders) | 0 (0) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 5 (5) | 1 (1)
ULCER, GI / STOMA (Gastrointestinal disorders) | 0 (0) | 1 (1)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 2 (2) | 2 (2)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 1 (1) | 0 (0)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VISION-BLURRED VISION (Eye disorders) | 2 (2) | 1 (1)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
VOMITING (Gastrointestinal disorders) | 4 (5) | 6 (6)
WEIGHT GAIN (General disorders) | 2 (2) | 0 (0)
WEIGHT LOSS (General disorders) | 2 (3) | 9 (11)

LIMITATIONS AND CAVEATS:
The primary object analysis was under powered. The sample size calculation determined 34 subjects per arm, however the actual primary objective analysis was based on 31 subjects per arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No